CLINICAL TRIAL: NCT01344915
Title: RESTRICTED VS. FREE KNEE RANGE OF MOTION FOR PRIMARY TRAUMATIC PATELLAR DISLOCATION: A PROSPECTIVE RANDOMIZED STUDY
Brief Title: Restricted vs. Free Knee Range Of Motion For Primary Traumatic Patellar Dislocation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Department of Orthopaedic Surgery, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PATRCTFIN
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2005-01

CONDITIONS: Patellar Dislocation
Keywords: Patella; Knee; Brace
MeSH Terms: conditions — Patellar Dislocation; Patella Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Knee brace (Active Comparator)
  Interventions: Procedure: Locked knee brace
- Locked knee brace (Active Comparator)
  Interventions: Procedure: Locked knee brace

INTERVENTIONS:
Procedure: Locked knee brace
  Arms: Knee brace
Procedure: Locked knee brace
  Arms: Locked knee brace

SUMMARY:
Knee immobilization in near extension has been proposed as a nonoperative treatment for primary traumatic patellar dislocation, although there exist no prospective studies regarding the method of immobilization. The objective of this prospective randomized study was to compare the clinical outcome after nonoperative treatment with restricted vs. free range of motion (ROM) for primary traumatic patellar dislocation.

ELIGIBILITY:
Inclusion Criteria:

* A primary (first-time) patellar dislocation verified by clinical examination
* Signs of patellar dislocation in MRI

Exclusion Criteria:

* anyone with previous patellar instability
* osteochondral fracture requiring surgery
* associated knee injuries

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2005-12; Primary Completion 2007-01 (Actual); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Patellar redislocation
  The number of patients with patellar redislocation after initial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Petri J Sillanpää, MD PhD, Principal Investigator — Tampere University Hospital, Department of Orthopaedic Surgery
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Honkonen EE, Sillanpaa PJ, Reito A, Maenpaa H, Mattila VM. A Randomized Controlled Trial Comparing a Patella-Stabilizing, Motion-Restricting Knee Brace Versus a Neoprene Nonhinged Knee Brace After a First-Time Traumatic Patellar Dislocation. Am J Sports Med. 2022 Jun;50(7):1867-1875. doi: 10.1177/03635465221090644. Epub 2022 Apr 19. PMID 35438588